CLINICAL TRIAL: NCT00472836
Title: A Phase 1, Open-Label, Parallel Group, Multiple-Dose Study To Evaluate The Pharmacokinetics, Safety And Toleration Of CP-945,598 Administered To Subjects With Severely Impaired And Normal Renal Function
Brief Title: Study Examining The Effect Of Renal Impairment On Safety, Toleration And How The Body Processes An Experimental Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5351038
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2008-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal renal function (Experimental)
  Interventions: Drug: CP-945,598
- Severe renal impairment (Experimental)
  Interventions: Drug: CP-945,598

INTERVENTIONS:
Drug: CP-945,598 — Administration of CP-945,598 in subjects with normal renal function.
  Arms: Normal renal function
Drug: CP-945,598 — Administration of CP-945,598 in subjects with severe renal impairment.
  Arms: Severe renal impairment

SUMMARY:
CP-945,598 is eliminated following extensive metabolism. For some drugs, decreased renal (kidney) function can affect their elimination from the body via metabolism. This study will therefore compare the pharmacokinetics (time course of drug concentrations in the body), safety and tolerability of CP-945,598 in patients with severe renal impairment and healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normal Subjects: 1.Healthy. 2.Matched for age (± 5 yrs), weight (± 10 kg), and gender ratio (± 2 subjects per gender).
* Subjects with Renal Disease: 1. Severe impairment (Creatinine clearance <30 mL/min) 2. Stable renal disease:no change in the last 30 days. 3. Stable dose of medication and/or treatment. 4. Reasonably well-controlled type 1 and type 2 diabetics

Exclusion Criteria:

* All subjects: Non-prescribed use of drugs of abuse/ recreational drugs; recent treatment with experimental drugs or herbal experiments; EKG and blood pressure parameters falling outside of protocol-specified limits; history of regular alcohol or tobacco use exceeding protocol-specified limits
* Normal subjects: Medically important health conditions; recent use of prescription or non-prescription medications.
* Subjects with renal disease: Subjects requiring dialysis; certain chronic medical conditions; patients who have received renal transplant; severe and/or poorly controlled diabetes; Treatment with protocol-specified drugs that may alter the way the body absorbs or processes CP-945,598.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Measurement of drug and metabolite concentrations in serum from blood samples collected at various times over 24 hour dosing interval on Days 1 & 14, before daily dose on days 2, 5-7, 13, following stopping of drug treatment on days 15-18, 21, | 14 days
28, 35 | 14 days

SECONDARY OUTCOMES:
Vital signs (blood pressure, heart rate and respiratory rate) on days 1, 2, 7, and 14 | 14 days
ECGs on Days 1,7 and 14 | 14 days
Safety laboratory tests (Chemistry, hematology, urinalysis) on Days 2, 7, 14 and 35 | 14 days
Adverse event monitoring throughout duration of the study | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Miami, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351038&StudyName=Study%20Examining%20The%20Effect%20Of%20Renal%20Impairment%20On%20Safety%2C%20Toleration%20And%20How%20The%20Body%20Processes%20An%20Experimental%20Drug